CLINICAL TRIAL: NCT00952835
Title: Evaluation of Different Disease Control Indices in Children With Asthma and Rhinitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Collaborators: Azienda Ospedaliera Universitaria Policlinico (Other)
Responsible Party: Principal Investigator, Boner Attilio, full professor, Universita di Verona
Other Study IDs: AOV-1716
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Asthma; Rhinitis
Keywords: Asthma; rhinitis; EIB; Exhaled Nitric oxide; lung function; vitamin d
MeSH Terms: conditions — Asthma; Rhinitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- asthma and rhinitis control
  Interventions: Other: regular treatment

INTERVENTIONS:
Other: regular treatment — regular treatment
  Other Names: asthma treatment

SUMMARY:
In this study will be consecutive enrolled children with asthma (classified according to GINA guidelines) and rhinitis (classified by ARIA guidelines); the investigators will research clinical personal and parental history regarding allergic diseases, exposition to passive smoking and interpretate hematochemical parameters markers of atopy. Skin Prick Tests will be performed. In this study the investigators will evaluate lung function parameters (spirometry with bronchial reversibility test and exercise induced bronchoconstriction, oscillometry, respiratory plethysmography, etc.), airway inflammatory indices such as exhaled nitric oxide at different flows, exhaled and nasal temperature, nasal cytology.

The aim of the study will be to evaluate possible correlation between these different parameters and clinical status of the patients.

DETAILED DESCRIPTION:
Each patients will be evaluated by spirometry and then he will undergo exercise challenge in order to evaluate exercise-induced bronchoconstriction as a marker of asthma control. The test of the challenge will be correlate with childhood Asthma control test score,levels of control (GINA classification)and the different markers of airway inflammation and atopy.

ELIGIBILITY:
Inclusion Criteria:

* patient with asthma and rhinitis

Exclusion Criteria:

* age <5 years
* chronic respiratory diseases

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: children with asthma and/or rhinitis visited at the outpatients clinic at the University of Verona will be invited to participate to the study
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Different Disease Control Indices in Children With Asthma and Rhinitis | Evaluation of Different Disease Control Indices in Children With Asthma and Rhinitis

CONTACTS AND LOCATIONS:
Overall Officials: Attilio Boner, MD, Principal Investigator — Universita di Verona
Locations (1):
- Pediatric department University of Verona, Verona, Verona, Italy

REFERENCES:
- [Derived] Chinellato I, Piazza M, Peroni D, Sandri M, Chiorazzo F, Boner AL, Piacentini G. Bronchial and alveolar nitric oxide in exercise-induced bronchoconstriction in asthmatic children. Clin Exp Allergy. 2012 Aug;42(8):1190-6. doi: 10.1111/j.1365-2222.2012.03973.x. PMID 22805466
- [Derived] Peroni DG, Cattazzo E, Chinellato I, Piazza M, Tezza G, Boner AL, Piacentini GL. Nasal mucosa temperature as a marker of disease in children with allergic rhinitis. Am J Rhinol Allergy. 2012 Jul-Aug;26(4):e115-8. doi: 10.2500/ajra.2012.26.3803. PMID 22801008